CLINICAL TRIAL: NCT00742560
Title: A Phase 1b/2, Multicenter, Open-label, Dose-escalation Study of Elotuzumab (Humanized Anti-CS1 Monoclonal IgG1 Antibody) in Combination With Lenalidomide and Dexamethasone in Subjects With Relapsed Multiple Myeloma
Brief Title: A Phase 1b/2, Dose-Escalation Study of Elotuzumab (Humanized Anti-CS1 Monoclonal IgG1 Antibody) in Relapsed Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HuLuc63-1703; 2007-006677-83 (EudraCT Number)
Record Dates: First submitted 2008-08-25; First posted 2008-08-27 (Estimated); Results first posted 2018-01-10 (Actual); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Hematologic Cancer
Keywords: Multiple Myeloma
MeSH Terms: conditions — Hematologic Neoplasms; Multiple Myeloma | interventions — elotuzumab; Lenalidomide; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Elotuzumab 5 mg/kg + Lenalidomide and Dexamethasone (Phase 1) (Experimental): Elotuzumab 5 mg/kg administered as an IV infusion in combination with lenalidomide 25 mg and dexamethasone 40 mg administered orally.
  Interventions: Biological: elotuzumab; Drug: lenalidomide; Drug: dexamethasone oral; Drug: dexamethasone injection
- Elotuzumab 10 mg/kg + Lenalidomide and Dexamethasone (Phase 1) (Experimental): Elotuzumab 10 mg/kg administered as an IV infusion in combination with lenalidomide 25 mg and dexamethasone 40 mg administered orally.
  Interventions: Biological: elotuzumab; Drug: lenalidomide; Drug: dexamethasone oral; Drug: dexamethasone injection
- Elotuzumab 20 mg/kg + Lenalidomide and Dexamethasone (Phase 1) (Experimental): Elotuzumab 20 mg/kg administered as an IV infusion in combination with lenalidomide 25 mg and dexamethasone 40 mg administered orally.
  Interventions: Biological: elotuzumab; Drug: lenalidomide; Drug: dexamethasone oral; Drug: dexamethasone injection
- Elotuzumab 10 mg/kg + Lenalidomide and Dexamethasone (Phase 2) (Experimental): Elotuzumab 10 mg/kg administered as an IV infusion in combination with lenalidomide 25 mg and dexamethasone 40 mg administered orally.
  Interventions: Biological: elotuzumab; Drug: lenalidomide; Drug: dexamethasone oral; Drug: dexamethasone injection
- Elotuzumab 20 mg/kg + Lenalidomide and Dexamethasone (Phase 2) (Experimental): Elotuzumab 20 mg/kg administered as an IV infusion in combination with lenalidomide 25 mg and dexamethasone 40 mg administered orally.
  Interventions: Biological: elotuzumab; Drug: lenalidomide; Drug: dexamethasone oral; Drug: dexamethasone injection

INTERVENTIONS:
Biological: elotuzumab — Humanized Anti-CS1 Monoclonal IgG1 Antibody (HuLuc63) administered as an intravenous infusion once a week during Cycles 1 and 2, and every other week beginning with Cycle 3.
  Other Names: HuLuc63
Drug: lenalidomide — Lenalidomide 25 mg administered orally once daily on Days 1 to 21 of each 28-day cycle
Drug: dexamethasone oral — Dexamethasone 40 mg administered orally once weekly; during weeks when elotuzumab is also administered, dexamethasone was administered as a split dose (28 mg orally and 8 mg intravenously)
Drug: dexamethasone injection — Dexamethasone 40 mg administered orally once weekly; during weeks when elotuzumab is also administered, dexamethasone was administered as a split dose (28 mg orally and 8 mg intravenously)

SUMMARY:
The purpose of this study is to evaluate the combination of elotuzumab, lenalidomide, and dexamethasone in subjects with relapsed multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older with a confirmed diagnosis of multiple myeloma (MM) and documentation of one to three prior therapies.
2. Confirmed evidence of disease progression from immediately prior MM therapy or refractory to the immediately prior treatment.
3. Measurable monoclonal (M-) protein component in serum (≥ 0.5 g/dL) and/or urine (if present), (≥ 0.2 g excreted in a 24 hour collection sample). Subjects with free light chain only disease are excluded.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 2.
5. Creatinine clearance ≥ 50 mL/min measured by Cockcroft-Gault method.
6. Hematologic parameters defined by:

   * Absolute neutrophil count >1000 cells/mm^3 without growth factors for 7 days.
   * Platelets ≥ 75,000 cells/mm^3 (75 × 10^9/L), without platelet transfusion, within 72 hours of screening evaluation.
   * Hemoglobin ≥ 8 g/dL without red blood cell transfusion within 72 hours of screening.
7. Alanine aminotransferase (ALT) AND aspartate aminotransferase (AST) < 3 × upper limit of normal.
8. Total bilirubin < 2 × upper limit of normal, direct bilirubin < 2.0 mg/dL.
9. Negative urine pregnancy test in women of childbearing potential at screening and prior to prescribing lenalidomide. Females of childbearing potential (FCBP) must either commit to continued abstinence from heterosexual intercourse or begin acceptable methods of birth control for 28 days prior to prescribing lenalidomide. Men must agree to use a latex condom during sexual contact with FCBP even if they have had a successful vasectomy, and must agree not to donate semen during study drug therapy and for a period of time after therapy.
10. Able to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (in accordance with national and local subject's privacy regulations).
11. Able to take aspirin daily as prophylactic anticoagulation therapy (subjects intolerant to aspirin may use warfarin or low-molecular-weight heparin).

Exclusion Criteria:

1. Prior malignancy, except for adequately treated basal cell or squamous cell skin cancer, in-situ cervical cancer, or other cancer from which the subject has been disease-free for at least 2 years.
2. Active or prior plasma cell leukemia (defined as either 20% of peripheral WBC comprised of plasma/CD138+ cells or an absolute count of 2 x 10^9/L).
3. Uncontrolled medical problems such as diabetes mellitus, coronary artery disease, hypertension, unstable angina, arrhythmias, pulmonary disease, and symptomatic heart failure.
4. Solitary bone or solitary extramedullary plasmacytoma as the only evidence of plasma cell dyscrasia.
5. Treatment with any investigational drug within 2 weeks or 3 half lives (whichever is longer) of the first dose of elotuzumab.
6. Use of corticosteroids, thalidomide, bortezomib, or cytotoxic chemotherapy within 2 weeks of the first dose of elotuzumab except for steroids with little or no systemic absorption (ie, topical or inhaled steroids).
7. Prior lenalidomide therapy.
8. Prior peripheral stem-cell transplant within 12 weeks of the first dose of elotuzumab.
9. Treatment with nitrosoureas, such as carmustine (BiCNU), nitrogen mustard agents, or melphalan, within 6 weeks of first dose of elotuzumab.
10. Neuropathy ≥ Grade 3 or painful neuropathy ≥ Grade 2 (National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] v3.0).
11. Known active infections requiring IV antibiotic, antiviral, or antifungal therapy.
12. Hypersensitivity to recombinant proteins or excipients in elotuzumab, lenalidomide, or dexamethasone.
13. Female subjects who are pregnant or breastfeeding.
14. Subjects with serum calcium (corrected for albumin) ≥ 12 mg/dL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2008-08; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc, Study Director — AbbVie

REFERENCES:
- [Derived] Richardson PG, Jagannath S, Moreau P, Jakubowiak AJ, Raab MS, Facon T, Vij R, White D, Reece DE, Benboubker L, Zonder J, Tsao LC, Anderson KC, Bleickardt E, Singhal AK, Lonial S; 1703 study investigators. Elotuzumab in combination with lenalidomide and dexamethasone in patients with relapsed multiple myeloma: final phase 2 results from the randomised, open-label, phase 1b-2 dose-escalation study. Lancet Haematol. 2015 Dec;2(12):e516-27. doi: 10.1016/S2352-3026(15)00197-0. Epub 2015 Nov 16. PMID 26686406

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 101 participants were randomized (intent-to-treat [ITT] population); 1 subject did not receive study drug and is excluded from the analyses.
Period: Overall Study
Arm/Group | Elotuzumab 5 mg/kg + Lenalidomide and Dexamethasone (Phase 1) | Elotuzumab 10 mg/kg + Lenalidomide and Dexamethasone (Phase 1) | Elotuzumab 20 mg/kg + Lenalidomide and Dexamethasone (Phase 1) | Elotuzumab 10 mg/kg + Lenalidomide and Dexamethasone (Phase 2) | Elotuzumab 20 mg/kg + Lenalidomide and Dexamethasone (Phase 2)
Started (Safety population: all randomized participants who received at least 1 dose of study drug) | 3 | 3 | 22 | 36 | 37
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 22 | 36 | 37
Not completed — Adverse Event | 0 | 0 | 1 | 1 | 1
Not completed — Death | 0 | 2 | 0 | 2 | 3
Not completed — Subject's Decision | 1 | 0 | 2 | 3 | 3
Not completed — Investigator's Decision | 0 | 0 | 4 | 1 | 0
Not completed — Disease Progression | 1 | 0 | 5 | 17 | 16
Not completed — New Multiple Myeloma Therapy | 1 | 0 | 2 | 3 | 4
Not completed — Other | 0 | 1 | 8 | 9 | 9
Not completed — MIssing | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population: all randomized participants who received at least 1 dose of study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | Elotuzumab 5 mg/kg + Lenalidomide and Dexamethasone (Phase 1) | Elotuzumab 10 mg/kg + Lenalidomide and Dexamethasone (Phase 1) | Elotuzumab 20 mg/kg + Lenalidomide and Dexamethasone (Phase 1) | Elotuzumab 10 mg/kg + Lenalidomide and Dexamethasone (Phase 2) | Elotuzumab 20 mg/kg + Lenalidomide and Dexamethasone (Phase 2) | Total
Number analyzed (Participants) | 3 | 3 | 22 | 36 | 37 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.3 (7.23) | 64.7 (6.94) | 59.3 (10.87) | 60.6 (9.70) | 63.3 (9.76) | 61.7 (9.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 10 | 19 | 24 | 56
  Male | 1 | 2 | 12 | 17 | 13 | 45

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Elotuzumab in Combination With Lenalidomide and Dexamethasone (Phase 1)
Description: MTD was determined by testing increasing doses up to 20 mg/kg once daily dose escalation cohorts 1 to 3 with 3 patients each. MTD reflects highest dose of drug that did not cause an unacceptable side effect (dose limiting toxicity [DLT]) in more than 30% of patients; e.g., hematologic toxicities like Common Toxicity Criteria for Adverse Events (CTCAE) Grade 4 neutropenia in specific conditions, platelets < 10,000 cells/mm^3 that do not recover to 25,000 cells/mm^3; and specific non-hematologic/biochemical toxicities CTCAE Grade 3 or 4 (except fatigue and Grade 3 infections); CTCAE version 3.0 were used.
Time Frame: 4 weeks
Population: All participants in the safety population (all randomized participants who received at least 1 dose of study drug) in the escalation cohorts (Elotuzumab 5 mg/kg + Lenalidomide and Dexamethasone [Phase 1]; Elotuzumab 10 mg/kg + Lenalidomide and Dexamethasone [Phase 1]; and Elotuzumab 20 mg/kg + Lenalidomide and Dexamethasone [Phase 1]).
Measure: Number; unit: mg/kg
Groups:
- Phase 1 Elotuzumab + Lenalidomide and Dexamethasone: Elotuzumab (5, 10, or 20 mg/kg) administered as an IV infusion in combination with lenalidomide 25 mg and dexamethasone 40 mg administered orally.
Arm/Group | Phase 1 Elotuzumab + Lenalidomide and Dexamethasone
Number analyzed (Participants) | 28
mg/kg | 20

2. Primary Outcome: Objective Response Rate (ORR) According to the International Myeloma Working Group Uniform Response Criteria (Phase 2)
Description: ORR: Percentage of participants with confirmed complete response (CR; negative immunofixation on the serum and urine, disappearance of any soft tissue plasmacytomas, and ≤5% plasma cells in bone marrow), partial response (PR; ≥50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by ≥90% or to ≤200 mg per 24 hour; if serum and urine M-protein are unmeasurable, a ≥50% decrease in the difference between involved and uninvolved free light chain (FLC] levels is required in place of the M-protein criteria; if serum and urine M-protein are unmeasurable, and serum FLC is also unmeasurable, a ≥50% reduction in plasma cells is required in place of M-protein, provided baseline bone marrow plasma cell percentage was ≥30%; and, if present at baseline, a ≥50% reduction in the size of soft tissue plasmacytomas), very good PR (VGPR; normal FLC ratio and absence of clonal cells in bone marrow by immunohistochemistry or immunofluorescence), or stringent CR (sCR; CR plus VGPR).
Time Frame: From date of randomization until 60 days following the last infusion (or before initiation of new therapy), up to 101 months
Population: Safety population: All randomized participants who received at least 1 dose of study drug
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Total (Phase 2): Elotuzumab (10 or 20 mg/kg) administered as an IV infusion in combination with lenalidomide 25 mg and dexamethasone 40 mg administered orally.
Arm/Group | Elotuzumab 10 mg/kg + Lenalidomide and Dexamethasone (Phase 2) | Elotuzumab 20 mg/kg + Lenalidomide and Dexamethasone (Phase 2) | Total (Phase 2)
Number analyzed (Participants) | 36 | 37 | 73
percentage of participants | 91.7 [77.5 to 98.2] | 75.7 [58.8 to 88.2] | 83.6 [73.0 to 91.2]

3. Secondary Outcome: Objective Response Rate (ORR) According to the International Myeloma Working Group Uniform Response Criteria (Phase 1)
Description: as for outcome 2
Time Frame: From first dose of elotuzumab until 60 days following the last infusion (or before initiation of new therapy), up to 100.5 months
Population: Safety population: All randomized participants who received at least 1 dose of study drug
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Total (Phase 1): Elotuzumab (5, 10, or 20 mg/kg) administered as an IV infusion in combination with lenalidomide 25 mg and dexamethasone 40 mg administered orally.
Arm/Group | Elotuzumab 5 mg/kg + Lenalidomide and Dexamethasone (Phase 1) | Elotuzumab 10 mg/kg + Lenalidomide and Dexamethasone (Phase 1) | Elotuzumab 20 mg/kg + Lenalidomide and Dexamethasone (Phase 1) | Total (Phase 1)
Number analyzed (Participants) | 3 | 3 | 22 | 28
percentage of participants | 100 [29.2 to 100.0] | 100 [29.2 to 100.0] | 77.3 [54.6 to 92.2] | 82.1 [63.1 to 93.9]

4. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. The investigator assessed the relationship of each event to the use of study drug as either definitely related, probably related, possibly related or unrelated. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the subject and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent events (TEAEs/TESAEs) are defined as any event that began or worsened in severity after the first dose of study drug. For more details on adverse events please see the Adverse Event section.
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from first dose of study drug until 60 days after the last dose of study drug (up to 95 months)
Population: Safety population: All randomized participants who received at least 1 dose of study drug
Measure: Number; unit: participants
Arm/Group | Elotuzumab 5 mg/kg + Lenalidomide and Dexamethasone (Phase 1) | Elotuzumab 10 mg/kg + Lenalidomide and Dexamethasone (Phase 1) | Elotuzumab 20 mg/kg + Lenalidomide and Dexamethasone (Phase 1) | Elotuzumab 10 mg/kg + Lenalidomide and Dexamethasone (Phase 2) | Elotuzumab 20 mg/kg + Lenalidomide and Dexamethasone (Phase 2)
Number analyzed (Participants) | 3 | 3 | 22 | 36 | 37
participants
  Any TEAE | 3 | 3 | 22 | 36 | 37
  Any TESAE | 0 | 3 | 12 | 21 | 21
  TEAEs ≥ Grade 3 | 2 | 3 | 19 | 32 | 25
  TEAEs related to study drug | 3 | 3 | 16 | 29 | 26
  TESAEs related to study drug | 0 | 0 | 2 | 2 | 5

5. Secondary Outcome: Number of Participants With Infusion Reactions
Description: During Phase 1, a list of 118 pre-defined MedDRA preferred terms that had been adjudicated to be clinically relevant to infusion reactions by a safety committee was used to search for TEAEs that could potentially be associated with an infusion reaction following elotuzumab administration. Examples of these terms included angioedema, bronchospasm, chills, flushing, pyrexia, rash and urticaria. During Phase 2, the method for capturing TEAEs associated with an infusion reaction was modified to include investigators' designation of AEs judged as clinically relevant infusion reactions. The number of participants infusion reactions are provided overall and by highest toxicity grade (CTCAE v 3.0).
Time Frame: Cycles 1 and 2: Days 1, 8, 15, and 22 (day of infusion of elotuzumab) and Days 2, 9, 16, and 23 (day following infusion); and Cycles 3 and greater: Days 1 and 15 (day of infusion) and Days 2 and 16 (day after infusion) (up to 95 months)
Population: Safety population: All randomized participants who received at least 1 dose of study drug
Measure: Number; unit: participants
Arm/Group | Elotuzumab 5 mg/kg + Lenalidomide and Dexamethasone (Phase 1) | Elotuzumab 10 mg/kg + Lenalidomide and Dexamethasone (Phase 1) | Elotuzumab 20 mg/kg + Lenalidomide and Dexamethasone (Phase 1) | Elotuzumab 10 mg/kg + Lenalidomide and Dexamethasone (Phase 2) | Elotuzumab 20 mg/kg + Lenalidomide and Dexamethasone (Phase 2)
Number analyzed (Participants) | 3 | 3 | 22 | 36 | 37
participants
  Any reaction | 2 | 3 | 20 | 5 | 3
  Grade 5 | 0 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 1 | 0 | 0
  Grade 3 | 0 | 0 | 2 | 1 | 0
  Grade 2 | 0 | 1 | 5 | 1 | 1
  Grade 1 | 2 | 2 | 12 | 3 | 2

6. Secondary Outcome: Mean Serum Concentrations of Elotuzumab During Cycle 1
Description: Blood samples were collected during Phase 1, Cycle 1, prior to elotuzumab infusion (time 0 hours) and 30 minutes (0.5 hours) and 4 hours post-infusion (Day 1), 30 minutes (0.5 hours) post-infusion (Day 8 and Day 15), or 30 minutes (0.5 hours), 2 hours, and 4 hours post-infusion (Day 15). Blood samples were collected during Phase 2, Cycle 1, prior to elotuzumab infusion (time 0 hours) and 30 minutes (0.5 hours), 2 hours, and 4 hours post-infusion (Day 1), 30 minutes (0.5 hours) and 2 hours post-infusion (Day 8 and Day 15), or 30 minutes (0.5 hours), 2 hours, and 4 hours post-infusion (Day 15). The samples were analyzed for the concentration of elotuzumab using validated analytical methods. Mean serum concentrations on Cycle 1, Days 1, 8, 15, and 22 (measured in μg/mL) are reported overall (across Phase 1 and Phase 2) by dose.
Time Frame: Cycle 1: Days 1 (pre-infusion and 0.5, 2 and 4 hours post-infusion), 8 (pre-infusion and 0.5 and 2 hours post-infusion), 15 (pre-infusion and 0.5 hours and 2 hours post-infusion), and 22 (pre-infusion and 0.5, 2, and 4 hours post-infusion)
Population: Safety population: All randomized participants who received at least 1 dose of study drug, with evaluable data at given time point.
Measure: Mean (Standard Deviation); unit: μg/mL
Groups:
- Elotuzumab 5 mg/kg + Lenalidomide and Dexamethasone: Elotuzumab 5 mg/kg administered as an IV infusion in combination with lenalidomide 25 mg and dexamethasone 40 mg administered orally in Phase 1.
- Elotuzumab 10 mg/kg + Lenalidomide and Dexamethasone: Elotuzumab 10 mg/kg administered as an IV infusion in combination with lenalidomide 25 mg and dexamethasone 40 mg administered orally in Phase 1 and Phase 2.
- Elotuzumab 20 mg/kg + Lenalidomide and Dexamethasone: Elotuzumab 20 mg/kg administered as an IV infusion in combination with lenalidomide 25 mg and dexamethasone 40 mg administered orally in Phase 1 and Phase 2.
Arm/Group | Elotuzumab 5 mg/kg + Lenalidomide and Dexamethasone | Elotuzumab 10 mg/kg + Lenalidomide and Dexamethasone | Elotuzumab 20 mg/kg + Lenalidomide and Dexamethasone
Number analyzed (Participants) | 3 | 39 | 58
μg/mL
  Day 1: 0 hours | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  Day 1: 0.5 hours: number analyzed (Participants) | 3 | 39 | 57
  Day 1: 0.5 hours | 78.48 (21.33) | 217.90 (99.31) | 434.20 (202.74)
  Day 1: 2 hours: number analyzed (Participants) | 0 | 36 | 43
  Day 1: 2 hours |  | 213.31 (91.30) | 388.58 (112.94)
  Day 1: 4 hours: number analyzed (Participants) | 3 | 3 | 12
  Day 1: 4 hours | 85.56 (23.54) | 251.34 (31.92) | 525.98 (188.46)
  Day 8: 0 hours: number analyzed (Participants) | 3 | 37 | 55
  Day 8: 0 hours | 32.44 (8.91) | 92.47 (61.16) | 168.55 (56.43)
  Day 8: 0.5 hours: number analyzed (Participants) | 3 | 22 | 44
  Day 8: 0.5 hours | 133.37 (40.87) | 281.53 (117.35) | 593.80 (192.70)
  Day 8: 2 hours: number analyzed (Participants) | 0 | 12 | 9
  Day 8: 2 hours |  | 268.35 (107.44) | 520.97 (207.28)
  Day 15: 0 hours: number analyzed (Participants) | 3 | 37 | 58
  Day 15: 0 hours | 49.84 (28.28) | 111.11 (56.36) | 298.82 (231.17)
  Day 15: 0.5 hours: number analyzed (Participants) | 3 | 36 | 55
  Day 15: 0.5 hours | 140.09 (32.28) | 282.29 (100.29) | 661.91 (251.08)
  Day 22: 0 hours: number analyzed (Participants) | 3 | 38 | 54
  Day 22: 0 hours | 61.93 (53.66) | 135.92 (106.83) | 308.02 (144.61)
  Day 22: 0.5 hours: number analyzed (Participants) | 3 | 38 | 54
  Day 22: 0.5 hours | 168.61 (59.31) | 310.03 (165.14) | 699.70 (230.41)
  Day 22: 2 hours: number analyzed (Participants) | 1 | 35 | 40
  Day 22: 2 hours | 268.53 (NA) — The estimated standard deviation of one sample is undefined | 298.85 (114.35) | 704.48 (234.98)
  Day 22: 4 hours: number analyzed (Participants) | 2 | 3 | 10
  Day 22: 4 hours | 128.94 (42.04) | 538.88 (195.35) | 981.16 (280.28)

7. Secondary Outcome: Maximum Serum Concentration (Cmax) of Elotuzumab
Description: The maximum plasma concentration (Cmax; measured in ng/mL) is the highest concentration that a drug achieves in the blood after administration in a dosing interval. The Cmax of elotuzumab was to be estimated using non-compartmental methods and data reported as the mean ± standard deviation. No noncompartmental pharmacokinetic parameters (e.g., AUC, CL, V, t 1/2) were estimated due to sparse serum concentration collections.
Time Frame: Cycle 1: Days 1, 8, and 15; Cycle 2: Days 1 and 22; Cycle 3 and beyond: Day 1
Population: No noncompartmental pharmacokinetic parameters (e.g., AUC, CL, V, t 1/2) were estimated (collected data not reliable due to assay limitations caused by sparse serum concentrations).
Arm/Group | Elotuzumab 5 mg/kg + Lenalidomide and Dexamethasone | Elotuzumab 10 mg/kg + Lenalidomide and Dexamethasone | Elotuzumab 20 mg/kg + Lenalidomide and Dexamethasone
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Area Under the Concentration-time Curve From 0 to Infinity (AUC0-inf) of Elotuzumab
Description: The area under the plasma concentration-time curve (AUC; measured in ng*hr/mL) is a method of measurement to determine the total exposure of a drug in blood plasma. The AUC24 of elotuzumab was to be estimated using non-compartmental methods and data reported as the mean ± standard deviation. No noncompartmental pharmacokinetic parameters (e.g., AUC, CL, V, t 1/2) were estimated due to sparse serum concentration collections.
Time Frame: Cycle 1: Days 1, 8, and 15; Cycle 2: Days 1 and 22; Cycle 3 and beyond: Day 1
Population: as for outcome 7
Arm/Group | Elotuzumab 5 mg/kg + Lenalidomide and Dexamethasone | Elotuzumab 10 mg/kg + Lenalidomide and Dexamethasone | Elotuzumab 20 mg/kg + Lenalidomide and Dexamethasone
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Systemic Clearance (CL) of Elotuzumab
Description: Systemic clearance (CL, measured in mL/kg/hr) is a measure of the efficiency with which a drug is irreversibly removed from the body. The CL of elotuzumab was to be estimated using non-compartmental methods and data reported as the mean ± standard deviation. No noncompartmental pharmacokinetic parameters (e.g., AUC, CL, V, t 1/2) were estimated due to sparse serum concentration collections.
Time Frame: Cycle 1: Days 1, 8, and 15; Cycle 2: Days 1 and 22; Cycle 3 and beyond: Day 1
Population: as for outcome 7
Arm/Group | Elotuzumab 5 mg/kg + Lenalidomide and Dexamethasone | Elotuzumab 10 mg/kg + Lenalidomide and Dexamethasone | Elotuzumab 20 mg/kg + Lenalidomide and Dexamethasone
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Volume of Distribution (V) of Elotuzumab
Description: Volume of distribution (V, measured in L/kg) is the hypothetical volume of body fluid that would be required to dissolve the amount of drug needed to achieve the same concentration in the blood. The V of elotuzumab was to be estimated using non-compartmental methods and data reported as the mean ± standard deviation. No noncompartmental pharmacokinetic parameters (e.g., AUC, CL, V, t 1/2) were estimated due to sparse serum concentration collections.
Time Frame: Cycle 1: Days 1, 8, and 15; Cycle 2: Days 1 and 22; Cycle 3 and beyond: Day 1
Population: as for outcome 7
Groups:
- Elotuzumab 5 mg/kg + Lenalidomide and Dexamethasone (Phase 1): Elotuzumab 5 mg/kg administered as an IV infusion in combination with lenalidomide 25 mg and dexamethasone 40 mg administered orally in Phase 1.
Arm/Group | Elotuzumab 5 mg/kg + Lenalidomide and Dexamethasone (Phase 1) | Elotuzumab 10 mg/kg + Lenalidomide and Dexamethasone | Elotuzumab 20 mg/kg + Lenalidomide and Dexamethasone
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Serum Half-life (t1/2) of Elotuzumab
Description: The serum half-life of a drug (t1/2, measured in hours) is the time necessary to reduce the plasma concentration by half. The t1/2 of elotuzumab was to be estimated using non-compartmental methods and data reported as the mean ± standard deviation. No noncompartmental pharmacokinetic parameters (e.g., AUC, CL, V, t 1/2) were estimated due to sparse serum concentration collections.
Time Frame: Cycle 1: Days 1, 8, and 15; Cycle 2: Days 1 and 22; Cycle 3 and beyond: Day 1
Population: as for outcome 7
Groups:
- Elotuzumab 5 mg/kg Administered as an IV Infusion in Combinati: Elotuzumab 10 mg/kg administered as an IV infusion in combination with lenalidomide 25 mg and dexamethasone 40 mg administered orally in Phase 1 and Phase 2.
Arm/Group | Elotuzumab 5 mg/kg + Lenalidomide and Dexamethasone | Elotuzumab 5 mg/kg Administered as an IV Infusion in Combinati | Elotuzumab 20 mg/kg + Lenalidomide and Dexamethasone
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Duration of Response
Description: Duration of response is defined as the time from the initial objective response to disease progression or death, whichever occurs first. The distribution of duration of response was estimated for each treatment group using Kaplan-Meier methodology. Point estimates and 95% CIs for the median for the duration of response distribution are provided.
Time Frame: From first dose of elotuzumab (phase 1) or randomization (phase 2) until 60 days following the last infusion (or before initiation of new therapy), up to 101 months
Population: Safety population: All randomized participants who received at least 1 dose of study drug
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Elotuzumab 5 mg/kg + Lenalidomide and Dexamethasone (Phase 1) | Elotuzumab 10 mg/kg + Lenalidomide and Dexamethasone (Phase 1) | Elotuzumab 20 mg/kg + Lenalidomide and Dexamethasone (Phase 1) | Total (Phase 1) | Elotuzumab 10 mg/kg + Lenalidomide and Dexamethasone (Phase 2) | Elotuzumab 20 mg/kg + Lenalidomide and Dexamethasone (Phase 2) | Total (Phase 2)
Number analyzed (Participants) | 3 | 3 | 22 | 28 | 36 | 37 | 73
months | 4.47 [1.45 to 4.47] | 9.92 [NA to NA] — NA=Not calculable due to insufficient response events | NA [NA to NA] — NA=Median was not reached (max value was 58.22) | NA [NA to NA] — NA=Median was not reached (max value was 58.22) | 34.83 [14.6 to NA] — NA=Not calculable due to insufficient response events | 29.01 [15.0 to NA] — NA=Not calculable due to insufficient response events | 29.24 [18.2 to NA] — NA=Not calculable due to insufficient response events

13. Secondary Outcome: Time to Progression (TTP)
Description: TTP is defined as the time from first dose (phase 1) or time from randomization (phase 2) to disease progression. The distribution of TTP was estimated for each treatment group using Kaplan-Meier methodology. Point estimates and 95% CIs for the median for the TTP distribution are provided.
Time Frame: as for outcome 12
Population: Safety population: All randomized participants who received at least 1 dose of study drug
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Elotuzumab 5 mg/kg + Lenalidomide and Dexamethasone (Phase 1) | Elotuzumab 10 mg/kg + Lenalidomide and Dexamethasone (Phase 1) | Elotuzumab 20 mg/kg + Lenalidomide and Dexamethasone (Phase 1) | Total (Phase 1) | Elotuzumab 10 mg/kg + Lenalidomide and Dexamethasone (Phase 2) | Elotuzumab 20 mg/kg + Lenalidomide and Dexamethasone (Phase 2) | Total (Phase 2)
Number analyzed (Participants) | 3 | 3 | 22 | 28 | 36 | 37 | 73
months | 6.08 [6.05 to 6.08] | 11.53 [NA to NA] — NA=Not calculable due to insufficient progression events | 52.93 [7.43 to NA] — NA=Not calculable due to insufficient progression events | 52.93 [7.43 to NA] — NA=Not calculable due to insufficient progression events | 32.49 [14.9 to NA] — NA=Not calculable due to insufficient progression events | 19.94 [12.9 to 35.7] | 28.16 [15.4 to 35.8]

14. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the time from first dose (phase 1) or time from randomization (phase 2) to disease progression or death. The distribution of PFS was estimated for each treatment group using Kaplan-Meier methodology. Point estimates and 95% CIs for the median for the PFS distribution are provided.
Time Frame: as for outcome 12
Population: Safety population: All randomized participants who received at least 1 dose of study drug
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Elotuzumab 10 mg/kg Administered as an IV Infusion in Combinat: Elotuzumab 20 mg/kg administered as an IV infusion in combination with lenalidomide 25 mg and dexamethasone 40 mg administered orally.
Arm/Group | Elotuzumab 5 mg/kg + Lenalidomide and Dexamethasone (Phase 1) | Elotuzumab 10 mg/kg + Lenalidomide and Dexamethasone (Phase 1) | Elotuzumab 20 mg/kg + Lenalidomide and Dexamethasone (Phase 1) | Total (Phase 1) | Elotuzumab 10 mg/kg + Lenalidomide and Dexamethasone (Phase 2) | Elotuzumab 10 mg/kg Administered as an IV Infusion in Combinat | Total (Phase 2)
Number analyzed (Participants) | 3 | 3 | 22 | 28 | 36 | 37 | 73
months | 6.08 [6.05 to 6.08] | 22.23 [11.5 to 32.9] | NA [NA to NA] — NA=Median was not reached (max value was 58.91) | 32.92 [7.43 to NA] — NA=Not calculable due to insufficient survival events | 32.49 [14.9 to NA] — NA=Not calculable due to insufficient survival events | 25.00 [14.0 to 35.7] | 28.62 [16.6 to 43.1]

15. Secondary Outcome: Percentage of Participants With Treatment-emergent Anti-elotuzumab Antibody (ADA)
Description: Treatment-emergent (post-dose) positive elotuzumab-specific ADA is differentiated from pre-existing (positive at the predose time point) positive elotuzumab-specific ADA. The percentage of participants with confirmed treatment-emergent ADA overall by dose is provided.
Time Frame: From screening through 60-day follow up period (up to 101 months)
Population: All participants who received at least one dose of study drug and with at least one evaluable post-dose sample.
Measure: Number; unit: percentage of participants
Groups:
- Elotuzumab 5 mg/kg + Lenalidomide and Dexamethasone: Elotuzumab 5 mg/kg administered as an IV infusion in combination with lenalidomide 25 mg and dexamethasone 40 mg administered orally.
- Elotuzumab 10 mg/kg + Lenalidomide and Dexamethasone: Elotuzumab 10 mg/kg administered as an IV infusion in combination with lenalidomide 25 mg and dexamethasone 40 mg administered orally.
- Elotuzumab 20 mg/kg + Lenalidomide and Dexamethasone: Elotuzumab 20 mg/kg administered as an IV infusion in combination with lenalidomide 25 mg and dexamethasone 40 mg administered orally.
Arm/Group | Elotuzumab 5 mg/kg + Lenalidomide and Dexamethasone | Elotuzumab 10 mg/kg + Lenalidomide and Dexamethasone | Elotuzumab 20 mg/kg + Lenalidomide and Dexamethasone
Number analyzed (Participants) | 3 | 39 | 57
percentage of participants | 0 | 6 | 5

16. Secondary Outcome: Plasma Cell Myeloma Cytogenetic Subtype
Description: Plasma cell myeloma cytogenetic subtype was assessed at the screening visit using standard karyotyping and/or fluorescence in situ hybridization. The number of participants in each cytogenetic risk category are provided: High Risk (International Staging System [ISS] stage II or III and t(4;14) or del(17p) abnormality); Standard Risk (not high or low risk); and Low Risk (ISS stage I or II and absence of t(4;14), del(17p) and 1q21 abnormalities AND age < 55).
Time Frame: Screening (up to 14 days prior to dosing)
Population: Safety population: All randomized participants who received at least 1 dose of study drug
Measure: Number; unit: participants
Arm/Group | Elotuzumab 5 mg/kg + Lenalidomide and Dexamethasone (Phase 1) | Elotuzumab 10 mg/kg + Lenalidomide and Dexamethasone (Phase 1) | Elotuzumab 20 mg/kg + Lenalidomide and Dexamethasone (Phase 1) | Elotuzumab 10 mg/kg + Lenalidomide and Dexamethasone (Phase 2) | Elotuzumab 20 mg/kg + Lenalidomide and Dexamethasone (Phase 2)
Number analyzed (Participants) | 3 | 3 | 22 | 36 | 37
participants
  High Risk | 1 | 0 | 0 | 1 | 3
  Standard Risk | 2 | 3 | 17 | 30 | 24
  Low Risk | 0 | 0 | 3 | 2 | 3
  Not Reported | 0 | 0 | 2 | 3 | 7

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from first dose of study drug until 60 days after the last dose of study drug (up to 95 months).
Description: TEAEs and TESAEs are defined as any adverse event or serious adverse event that begins or worsens in severity after initiation of study drug until 30 days after the last dose of study drug.
Arm/Group | Elotuzumab 5 mg/kg + Lenalidomide and Dexamethasone (Phase 1) | Elotuzumab 10 mg/kg + Lenalidomide and Dexamethasone (Phase 1) | Elotuzumab 20 mg/kg + Lenalidomide and Dexamethasone (Phase 1) | Elotuzumab 10 mg/kg + Lenalidomide and Dexamethasone (Phase 2) | Elotuzumab 20 mg/kg + Lenalidomide and Dexamethasone (Phase 2)
Serious Adverse Events (participants affected / at risk) | 0/3 | 3/3 | 12/22 | 21/36 | 21/37
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 22/22 | 36/36 | 37/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Elotuzumab 5 mg/kg + Lenalidomide and Dexamethasone (Phase 1) (N=3) | Elotuzumab 10 mg/kg + Lenalidomide and Dexamethasone (Phase 1) (N=3) | Elotuzumab 20 mg/kg + Lenalidomide and Dexamethasone (Phase 1) (N=22) | Elotuzumab 10 mg/kg + Lenalidomide and Dexamethasone (Phase 2) (N=36) | Elotuzumab 20 mg/kg + Lenalidomide and Dexamethasone (Phase 2) (N=37)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1 | 2
LYMPHOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
ANGINA PECTORIS (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 1 | 1 | 0 | 1
BRADYCARDIA (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
TACHYCARDIA (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
CONSTIPATION (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
DIVERTICULAR PERFORATION (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
GASTROINTESTINAL PERFORATION (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
HAEMATEMESIS (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
VARICES OESOPHAGEAL (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
VOMITING (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
CHEST PAIN (General disorders) | 0 | 0 | 1 | 0 | 1
MULTIPLE ORGAN DYSFUNCTION SYNDROME (General disorders) | 0 | 0 | 0 | 0 | 1
PYREXIA (General disorders) | 0 | 0 | 0 | 0 | 2
CHOLECYSTITIS (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
ANAPHYLACTIC REACTION (Immune system disorders) | 0 | 0 | 1 | 0 | 0
ASPERGILLUS INFECTION (Infections and infestations) | 0 | 0 | 1 | 0 | 0
BRONCHITIS (Infections and infestations) | 0 | 0 | 0 | 2 | 1
CELLULITIS (Infections and infestations) | 0 | 0 | 0 | 2 | 1
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0
H1N1 INFLUENZA (Infections and infestations) | 0 | 0 | 0 | 1 | 0
HERPES ZOSTER (Infections and infestations) | 0 | 0 | 0 | 1 | 0
INFLUENZA (Infections and infestations) | 0 | 0 | 0 | 1 | 0
LOCALISED INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 0
LUNG INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 1
MENINGITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1
PNEUMONIA (Infections and infestations) | 0 | 0 | 1 | 4 | 5
PNEUMONIA KLEBSIELLA (Infections and infestations) | 0 | 0 | 0 | 0 | 1
PNEUMONIA VIRAL (Infections and infestations) | 0 | 0 | 0 | 1 | 0
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 0
PYELONEPHRITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1
SEPSIS (Infections and infestations) | 0 | 0 | 1 | 3 | 2
URINARY TRACT INFECTION (Infections and infestations) | 0 | 0 | 1 | 0 | 0
VISCERAL LEISHMANIASIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1
GASTROENTERITIS RADIATION (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
ELECTROLYTE IMBALANCE (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
BLADDER TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
LOBULAR BREAST CARCINOMA IN SITU (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
MYELODYSPLASTIC SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
GENERALISED TONIC-CLONIC SEIZURE (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
SYNCOPE (Nervous system disorders) | 0 | 0 | 0 | 2 | 0
TRANSIENT GLOBAL AMNESIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
CONFUSIONAL STATE (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0
RENAL COLIC (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
RENAL FAILURE (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
PROSTATITIS (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 0
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1
STRIDOR (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
RASH (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
ACCELERATED HYPERTENSION (Vascular disorders) | 0 | 0 | 0 | 1 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 0 | 1 | 0 | 1
PHLEBITIS (Vascular disorders) | 0 | 0 | 0 | 0 | 1
PHLEBITIS SUPERFICIAL (Vascular disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Elotuzumab 5 mg/kg + Lenalidomide and Dexamethasone (Phase 1) (N=3) | Elotuzumab 10 mg/kg + Lenalidomide and Dexamethasone (Phase 1) (N=3) | Elotuzumab 20 mg/kg + Lenalidomide and Dexamethasone (Phase 1) (N=22) | Elotuzumab 10 mg/kg + Lenalidomide and Dexamethasone (Phase 2) (N=36) | Elotuzumab 20 mg/kg + Lenalidomide and Dexamethasone (Phase 2) (N=37)
ANAEMIA (Blood and lymphatic system disorders) | 2 | 2 | 10 | 17 | 13
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 1 | 1 | 2 | 3
HAEMOGLOBINAEMIA (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
INCREASED TENDENCY TO BRUISE (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0
LEUKOPENIA (Blood and lymphatic system disorders) | 1 | 1 | 2 | 8 | 6
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 2
LYMPHOPENIA (Blood and lymphatic system disorders) | 0 | 1 | 1 | 12 | 8
NEUTROPENIA (Blood and lymphatic system disorders) | 2 | 3 | 7 | 12 | 9
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 3
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 | 2 | 5 | 12 | 10
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 1 | 1 | 1 | 3
PALPITATIONS (Cardiac disorders) | 0 | 0 | 2 | 2 | 2
HYPOACUSIS (Ear and labyrinth disorders) | 0 | 0 | 1 | 1 | 3
TINNITUS (Ear and labyrinth disorders) | 1 | 0 | 1 | 0 | 0
VERTIGO (Ear and labyrinth disorders) | 1 | 0 | 0 | 3 | 3
CATARACT (Eye disorders) | 0 | 0 | 2 | 4 | 6
DRY EYE (Eye disorders) | 0 | 0 | 1 | 0 | 2
EYE IRRITATION (Eye disorders) | 0 | 0 | 1 | 3 | 3
OCULAR HYPERAEMIA (Eye disorders) | 0 | 0 | 0 | 1 | 3
VISION BLURRED (Eye disorders) | 0 | 0 | 4 | 9 | 5
VISUAL ACUITY REDUCED (Eye disorders) | 0 | 0 | 0 | 3 | 1
VITREOUS FLOATERS (Eye disorders) | 0 | 0 | 1 | 0 | 2
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 | 0 | 1 | 4 | 2
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 1 | 7 | 7
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 0 | 0 | 5 | 4
CONSTIPATION (Gastrointestinal disorders) | 1 | 2 | 11 | 18 | 19
DIARRHOEA (Gastrointestinal disorders) | 1 | 2 | 14 | 24 | 25
DIVERTICULAR PERFORATION (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
DRY MOUTH (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 2
DYSPEPSIA (Gastrointestinal disorders) | 0 | 0 | 1 | 8 | 2
FLATULENCE (Gastrointestinal disorders) | 0 | 0 | 2 | 2 | 1
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
GASTROINTESTINAL MOTILITY DISORDER (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
GASTROINTESTINAL PERFORATION (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 | 0 | 1 | 3 | 4
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0
HAEMORRHOIDS (Gastrointestinal disorders) | 0 | 1 | 2 | 2 | 1
NAUSEA (Gastrointestinal disorders) | 0 | 3 | 11 | 18 | 17
PARAESTHESIA ORAL (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0
STOMATITIS (Gastrointestinal disorders) | 0 | 1 | 1 | 3 | 1
TOOTH DISORDER (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
TOOTHACHE (Gastrointestinal disorders) | 0 | 0 | 2 | 3 | 0
VOMITING (Gastrointestinal disorders) | 0 | 0 | 6 | 11 | 6
ASTHENIA (General disorders) | 0 | 1 | 6 | 7 | 12
CHEST DISCOMFORT (General disorders) | 0 | 0 | 1 | 1 | 2
CHEST PAIN (General disorders) | 0 | 0 | 1 | 0 | 3
CHILLS (General disorders) | 2 | 2 | 1 | 6 | 2
FATIGUE (General disorders) | 1 | 2 | 15 | 24 | 18
FEELING HOT (General disorders) | 0 | 0 | 0 | 2 | 0
GAIT DISTURBANCE (General disorders) | 0 | 0 | 1 | 2 | 2
INFLAMMATION (General disorders) | 0 | 0 | 0 | 2 | 0
INFLUENZA LIKE ILLNESS (General disorders) | 0 | 0 | 2 | 2 | 0
IRRITABILITY (General disorders) | 0 | 0 | 0 | 2 | 1
NON-CARDIAC CHEST PAIN (General disorders) | 0 | 0 | 1 | 5 | 2
OEDEMA (General disorders) | 0 | 0 | 0 | 5 | 1
OEDEMA PERIPHERAL (General disorders) | 0 | 1 | 6 | 14 | 9
PAIN (General disorders) | 0 | 0 | 4 | 1 | 5
PERIPHERAL SWELLING (General disorders) | 0 | 0 | 2 | 5 | 7
PYREXIA (General disorders) | 0 | 0 | 10 | 14 | 17
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 0 | 0 | 1 | 2 | 0
DRUG HYPERSENSITIVITY (Immune system disorders) | 0 | 0 | 0 | 2 | 1
SEASONAL ALLERGY (Immune system disorders) | 0 | 1 | 1 | 3 | 0
BRONCHITIS (Infections and infestations) | 0 | 0 | 5 | 8 | 10
CELLULITIS (Infections and infestations) | 0 | 0 | 0 | 4 | 4
CONJUNCTIVITIS (Infections and infestations) | 0 | 0 | 4 | 1 | 2
EAR INFECTION (Infections and infestations) | 0 | 0 | 0 | 2 | 0
FUNGAL INFECTION (Infections and infestations) | 0 | 1 | 0 | 1 | 0
GASTROENTERITIS (Infections and infestations) | 0 | 0 | 0 | 2 | 3
GASTROENTERITIS VIRAL (Infections and infestations) | 0 | 0 | 1 | 2 | 0
GINGIVITIS (Infections and infestations) | 0 | 0 | 2 | 1 | 0
HERPES ZOSTER (Infections and infestations) | 0 | 0 | 0 | 4 | 0
INFLUENZA (Infections and infestations) | 0 | 0 | 1 | 8 | 3
LOCALISED INFECTION (Infections and infestations) | 0 | 0 | 1 | 2 | 2
LUNG INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 3
NASOPHARYNGITIS (Infections and infestations) | 0 | 0 | 3 | 10 | 9
ORAL CANDIDIASIS (Infections and infestations) | 0 | 1 | 1 | 1 | 5
ORAL HERPES (Infections and infestations) | 0 | 0 | 0 | 2 | 1
PHARYNGITIS (Infections and infestations) | 0 | 0 | 0 | 1 | 2
PNEUMONIA (Infections and infestations) | 0 | 0 | 4 | 7 | 9
PNEUMONIA VIRAL (Infections and infestations) | 0 | 0 | 0 | 2 | 0
RHINITIS (Infections and infestations) | 1 | 0 | 1 | 5 | 8
SEPSIS (Infections and infestations) | 0 | 0 | 1 | 3 | 2
SINUSITIS (Infections and infestations) | 1 | 0 | 3 | 5 | 3
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1 | 7 | 19 | 15
UPPER RESPIRATORY TRACT INFECTION BACTERIAL (Infections and infestations) | 0 | 1 | 0 | 0 | 0
URINARY TRACT INFECTION (Infections and infestations) | 0 | 0 | 4 | 6 | 5
VIRAL INFECTION (Infections and infestations) | 0 | 1 | 1 | 0 | 0
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 1 | 0 | 2
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2
CONTUSION (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 4 | 4
FALL (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 5 | 4
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
SKIN ABRASION (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 2
STOMA SITE PAIN (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
SUNBURN (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 2 | 0
ACTIVATED PARTIAL THROMBOPLASTIN TIME PROLONGED (Investigations) | 0 | 0 | 0 | 2 | 1
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 0 | 1 | 5 | 4
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 0 | 0 | 3 | 4
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 | 0 | 2 | 3 | 1
BLOOD BICARBONATE DECREASED (Investigations) | 0 | 0 | 0 | 7 | 4
BLOOD CREATININE INCREASED (Investigations) | 0 | 0 | 2 | 5 | 4
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 0 | 0 | 0 | 4 | 1
BLOOD MAGNESIUM DECREASED (Investigations) | 0 | 0 | 1 | 2 | 0
BLOOD PHOSPHORUS DECREASED (Investigations) | 0 | 1 | 1 | 0 | 0
BLOOD POTASSIUM DECREASED (Investigations) | 0 | 1 | 1 | 0 | 0
BLOOD UREA INCREASED (Investigations) | 0 | 0 | 0 | 2 | 2
CARDIAC MURMUR (Investigations) | 0 | 0 | 0 | 3 | 1
EJECTION FRACTION DECREASED (Investigations) | 0 | 0 | 0 | 2 | 0
IMMUNOGLOBULINS DECREASED (Investigations) | 0 | 1 | 0 | 0 | 0
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 0 | 0 | 0 | 3 | 1
NEUTROPHIL COUNT INCREASED (Investigations) | 0 | 0 | 0 | 3 | 1
PROTEIN TOTAL INCREASED (Investigations) | 0 | 0 | 0 | 2 | 0
PROTHROMBIN TIME PROLONGED (Investigations) | 0 | 0 | 0 | 2 | 1
WEIGHT DECREASED (Investigations) | 0 | 0 | 3 | 7 | 4
WEIGHT INCREASED (Investigations) | 0 | 0 | 2 | 1 | 3
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 0 | 0 | 1 | 2 | 2
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 | 0 | 3 | 10 | 8
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 0 | 1 | 3 | 2
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 2
GOUT (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 2
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 3
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 3 | 9 | 12
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1 | 3 | 1
HYPERNATRAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 0
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 5 | 3
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 3
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 6 | 7 | 7
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 2
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1 | 3 | 2
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 5
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 3
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 2 | 7 | 12 | 8
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 7 | 17 | 14
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 4 | 8
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 | 1 | 10 | 22 | 23
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 1
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 5 | 4 | 3
MUSCULOSKELETAL DISCOMFORT (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 6 | 4
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 6 | 1
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 4 | 3
OSTEONECROSIS OF JAW (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 1 | 5 | 10 | 13
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 1
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 2
AMNESIA (Nervous system disorders) | 0 | 0 | 1 | 0 | 2
BALANCE DISORDER (Nervous system disorders) | 1 | 0 | 0 | 1 | 1
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 0 | 0 | 2 | 0 | 0
DISTURBANCE IN ATTENTION (Nervous system disorders) | 0 | 0 | 2 | 0 | 0
DIZZINESS (Nervous system disorders) | 0 | 0 | 4 | 12 | 7
DYSGEUSIA (Nervous system disorders) | 0 | 0 | 2 | 9 | 6
HEADACHE (Nervous system disorders) | 1 | 0 | 5 | 14 | 7
HYPOAESTHESIA (Nervous system disorders) | 0 | 0 | 1 | 5 | 3
HYPOGEUSIA (Nervous system disorders) | 0 | 0 | 0 | 2 | 0
MEMORY IMPAIRMENT (Nervous system disorders) | 0 | 0 | 2 | 2 | 2
NEURALGIA (Nervous system disorders) | 0 | 0 | 0 | 2 | 1
NEUROPATHY PERIPHERAL (Nervous system disorders) | 0 | 0 | 7 | 8 | 7
PARAESTHESIA (Nervous system disorders) | 1 | 0 | 3 | 6 | 3
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 0 | 0 | 1 | 3 | 5
PSYCHOMOTOR HYPERACTIVITY (Nervous system disorders) | 0 | 0 | 0 | 3 | 0
SCIATICA (Nervous system disorders) | 0 | 0 | 0 | 2 | 0
SINUS HEADACHE (Nervous system disorders) | 0 | 0 | 1 | 3 | 1
SOMNOLENCE (Nervous system disorders) | 0 | 0 | 0 | 2 | 1
SYNCOPE (Nervous system disorders) | 0 | 0 | 1 | 6 | 1
TREMOR (Nervous system disorders) | 0 | 0 | 0 | 3 | 5
AGGRESSION (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0
ANXIETY (Psychiatric disorders) | 0 | 0 | 4 | 5 | 1
CONFUSIONAL STATE (Psychiatric disorders) | 0 | 0 | 0 | 1 | 3
DEPRESSED MOOD (Psychiatric disorders) | 0 | 0 | 0 | 2 | 1
DEPRESSION (Psychiatric disorders) | 1 | 0 | 2 | 4 | 3
INSOMNIA (Psychiatric disorders) | 2 | 1 | 7 | 10 | 15
MOOD SWINGS (Psychiatric disorders) | 0 | 0 | 2 | 1 | 2
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0
DYSURIA (Renal and urinary disorders) | 0 | 0 | 1 | 4 | 2
HAEMATURIA (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 2
POLLAKIURIA (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2
RENAL FAILURE (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 2
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 3
VULVOVAGINAL PRURITUS (Reproductive system and breast disorders) | 0 | 0 | 0 | 2 | 0
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 7 | 12 | 13
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 6 | 3
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 5 | 11 | 10
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 9 | 5
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 6 | 6
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 3
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 2
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2 | 5
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 5 | 4
PARANASAL SINUS HYPERSECRETION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 1
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 5 | 2
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 2
RALES (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 4 | 5
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 4 | 2
THROAT IRRITATION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 1
UPPER-AIRWAY COUGH SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2 | 1
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3 | 0
BLISTER (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1 | 1
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 3 | 3
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 3 | 4
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 4 | 5
INGROWING NAIL (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 8 | 10
PRURITUS (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 2 | 2
RASH (Skin and subcutaneous tissue disorders) | 1 | 1 | 3 | 9 | 9
RASH GENERALISED (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 2 | 2
RASH MACULAR (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 1
SCAB (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2
SKIN DISCOLOURATION (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2
SKIN LESION (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 1
URTICARIA (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 | 0 | 3 | 2 | 2
FLUSHING (Vascular disorders) | 0 | 0 | 1 | 4 | 2
HOT FLUSH (Vascular disorders) | 0 | 1 | 2 | 2 | 2
HYPERTENSION (Vascular disorders) | 0 | 0 | 2 | 2 | 2
HYPOTENSION (Vascular disorders) | 0 | 0 | 3 | 4 | 4
PHLEBITIS SUPERFICIAL (Vascular disorders) | 0 | 0 | 0 | 2 | 0
THROMBOPHLEBITIS SUPERFICIAL (Vascular disorders) | 0 | 0 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.